CLINICAL TRIAL: NCT05239026
Title: Treadmill Training With Concurrently Controlled Speed and Cadence in People With Parkinson's Disease
Brief Title: Treadmill Training in People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Feng Yang, PhD, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H22192
Record Dates: First submitted 2022-01-06; First posted 2022-02-14 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Training Group (Experimental): This arm will receive a single session treadmill training session in which both cadence and treadmill speed are controlled.
  Interventions: Behavioral: Advanced treadmill walking
- Traditional Training Group (Experimental): This arm will receive a single session treadmill training session in which only treadmill speed is controlled.
  Interventions: Behavioral: Traditional treadmill walking

INTERVENTIONS:
Behavioral: Advanced treadmill walking — Participants will walking on a treadmill for 6 5-minute Blocks. The cadence will be progressively reduced for the first 3 Blocks. Speed will progressively increase during Blocks 4-6 while cadence from Block 3 is maintained.
  Arms: Advanced Training Group
Behavioral: Traditional treadmill walking — Participants will walking on a treadmill for 6 5-minute Blocks. Participants will walk at self-selected cadence during Blocks 1-3. Speed will progressively increase during Blocks 4-6.
  Arms: Traditional Training Group

SUMMARY:
The study will explore if coupling speed and cadence during treadmill training elicit more benefits than controlling speed alone in individuals with Parkinson's disease.

DETAILED DESCRIPTION:
Impaired gait is prevalent and raises the fall risk in people with Parkinson's Disease (PwPD). Gait speed, step length, and cadence are three interrelated components of human gait, as speed is determined by step length and cadence. Auditory cues, such as metronomes, have been shown to aid training for PwPD. The purpose of this study is to examine if controlling cadence and speed improves overground gait parameters in PwPD better than only controlling speed. Two groups of PwPD will participate. Both groups will attend a single treadmill training session. Both groups will complete overground walking trials as a pre-test measurement. One group will receive treadmill training in which cadence, via a metronome, and speed are controlled, while only speed is controlled for the other group. Both groups will complete the same overground walking trials as a post-test measurements. The specific aim of this study is to determine the effects of metronome cues and gait speed versus gait speed alone treadmill training on spatiotemporal gait parameters when walking overground in PwPD.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English
* Between the ages of 18-89 years old
* Diagnosed with Parkinson's Disease
* Stage 1-3 based on the Hoehn and Yahr
* Able to walk overground more than 15m independently
* Able to walk on a treadmill for at least 15 minutes independently

Exclusion Criteria:

* Diagnosed with any uncontrolled cardiorespiratory or metabolic disease
* Experience any other known neurologic disorders that affect their ability to walk
* Diagnosed with any visual or communication disorders
* Suffered a lower extremity injury within the last 6 months

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Gait Speed Determined based on the Time Measured by A Stop Watch and the 10-meter Walking Distance at Post-intervention Assessment Which Is about One Hour Later Than the Baseline Test. | Baseline and post-intervention (about 1 hour following the baseline)
  Gait speed will be calculated as the 10-meter walking distance divided by the time used to cover this distance and reported in meters/second. A 10-meter walkway is valid and reliable as an assessment of gait speed. A stop watch is a valid and reliable way to measure the walking time.

SECONDARY OUTCOMES:
Change from Baseline in the Step Length Determined by the Vicon Motion Capture System at Post-intervention Assessment Which Is about One Hour Later Than the Baseline Test. | Baseline and post-intervention (about 1 hour following the baseline)
  Step length, in meters, will be measured using a 9-camera Vicon motion capture system as the anteroposterior distance between heel markers at initial contact during overground walking. The Vicon motion capture system is valid and reliable to measure human body movement.
Change from Baseline in the Step Cadence as Assessed by the Vicon Motion Capture System at Post-intervention Assessment Which Is about One Hour Later Than the Baseline Test. | Baseline and post-intervention (about 1 hour following the baseline)
  Step frequency is the number of steps taken during overground walking and reported as steps/min. The Vicon motion capture system is valid and reliable to counter the number of steps taken by a participant within a minute.
Change from Baseline in Dynamic Gait Stability Assessed by the Feasible Stability Region Theory at Post-intervention Assessment Which Is about One Hour Later Than the Baseline Test. | Baseline and post-intervention (about 1 hour following the baseline)
  Dynamic gait stability is a unitless metric and will be calculated based on the Feasible Stability Region theoretical framework. The Feasible Stability Region framework has been valid and broadly used to quantify dynamic gait stability.
Change from Baseline in Ground Reaction Force Assessed by Force Plates at Post-intervention Assessment Which Is about One Hour Later Than the Baseline Test. | Baseline and post-intervention (about 1 hour following the baseline)
  Ground reaction force will be be measured by two force plates (AMTI, MA) during overground walking and will be expressed in Newtons. AMTI force plates are valid and reliable to evaluate the ground reaction forces during human walking.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Yang, PhD, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No